CLINICAL TRIAL: NCT05633836
Title: Indocyanine Green FLUorescence-guided Surgery to Achieve MICROscopic Cytoreduction After Macroscopically Complete Cytoreductive Surgery in Patients With Epithelial Ovarian Cancer
Brief Title: MicroFluO: FLUorescence-guided Surgery for Ovarian Cancer
Acronym: MicroFluO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Site de Recherche Intégrée sur le Cancer - CAncer Research for PErsonalized Medicine (SIRIC-CARPEM), France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP220637; 2022-A00522-41 (Registry Identifier: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; fluorescence guided surgery; indocyanine green; cytoreductive surgery; peritoneal carcinomatosis
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluorescence guided surgery (Experimental): During exploratory laparoscopy or at the end of macroscopically complete cytoreductive surgery, indocyanine green fluorescence-guided surgery is performed to identify peritoneal carcinoma lesions not visible in white light
  Interventions: Procedure: Fluorescence guided surgery

INTERVENTIONS:
Procedure: Fluorescence guided surgery — During exploratory laparoscopy or at the end of macroscopically complete cytoreduction surgery, indocyanine green fluorescence-guided surgery is performed to identify peritoneal carcinoma lesions not visible in white light

SUMMARY:
Epithelial ovarian cancers (EOC) are discovered in 75% of cases at an advanced stage, marked by the presence of peritoneal carcinomatosis. It has been shown that one of the main prognostic factors is the achievement of a macroscopically complete cytoreductive surgery, i.e. without visible peritoneal metastasis at the end of the procedure. The prognosis of patients is inversely correlated to the tumor residue at the end of the procedure, and 60% of patients present a peritoneal recurrence within two years after the initial management. This suggests that microscopic peritoneal metastases may be present that are not eradicated by surgery and not controlled by systemic chemotherapy. Their presence could be involved in the mechanisms leading to the occurrence of peritoneal recurrence.

The MicroPCI protocol (NCT03754569), showed that microscopic peritoneal metastases were present at the end of macroscopically complete surgery of advanced-stage EOC in 98.14% of cases.This naturally lead to the question of the impact of microscopic cytoreduction on the prognosis of patients. Fluorescence detection of peritoneal metastases after intravenous injection of indocyanine green (ICG) and their resection have already been evaluated with promising results in digestive and ovarian carcinomas.

The objective of the MicroFluO protocol is to propose on the one hand a diagnostic time by fluorescence during the laparoscopic evaluation performed to define the resectability of the peritoneal carcinomatosis and also at the end of the macroscopically complete cytoreductive surgery to perform the biopsy of the fluorescent areas suspected of presenting residual microscopic peritoneal metastases.

Patients diagnosed with peritoneal carcinomatosis undergo exploratory laparoscopy, during which lesion mapping is performed to assess the resectability of the lesions. A biopsy is performed during this procedure to confirm the histological diagnosis. An initial fluorescence mapping will be performed at this diagnostic time.

Once cytoreductive surgery has been performed, intravenous injection of ICG is performed according to the manufacturer's recommendations. Peritoneal lesions emitting a fluorescent signal will be sampled. These samples will be studied in anatomopathology under the same conditions as the other surgical parts.

No increase in morbidity is expected in relation to this study. The number of specimens taken is dependent on the peritoneal tumor burden.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years of age.
* Presenting with an epithelial ovarian cancer
* Affiliated to a social security system
* Having received full information on the organization of the research and having given written consent.

Exclusion Criteria:

* Borderline ovarian tumor.
* Non French speaking patient.
* Patient under a legal protection measure (guardianship, curatorship, safeguard of justice).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Rate of microscopic metastases detected by fluorescence | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Hôpital européen Georges-Pompidou, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).